CLINICAL TRIAL: NCT05893446
Title: Essential Connections: How Improved Referrals From Hospital to Community Meal Provision Can Impact Malnutrition Outcomes in Older Adults
Brief Title: Essential Connections: Hospital to Community Impacting Malnutrition Outcomes in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academy of Nutrition and Dietetics (Other)
Collaborators: University of New Mexico (Other); Hartford Hospital (Other); Meals on Wheels Central Texas (Other)
Responsible Party: Principal Investigator, Alison L Steiber, Chief Science Officer, Academy of Nutrition and Dietetics
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 95INNU0045
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Malnutrition; Protein
MeSH Terms: conditions — Kwashiorkor | interventions — Meals

STUDY DESIGN:
Intervention Model Description: Patient enrollment and data collection will begin in year two. In year one, sites will have been randomized to the intervention condition within four sequence blocks on a staggered schedule. The stepped wedge cluster-randomized trial design will go through 5 periods with each period lasting for 7 months for a total of 35 months (year 2 through year 4). The goal of year two is for all sites to initiate the schedule to which they are randomly assigned. All participating sites will start in the control condition (usual process/care) in period 1. By the end of year two, we aim for sites to be within period 2. At this time, two sites will be implementing the intervention. Patients will be recruited and enrolled from acute care hospital sites in a rolling fashion across the entire study period (year 2 to year 4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Nutrition care by RDN, medical nutrition therapy -stepped wedge cluster-randomized trial design. Everyone gets the intervention so no arms. — RDNs in the community will provide MNT and meals for three months post discharge from the hospital
  Other Names: Meals

SUMMARY:
Meal provision organizations, whether they provide meals within the home or in congregate centers, provide an excellent opportunity to address malnutrition by providing nutrition care and meals to those who are most vulnerable. Data has shown that nutrition care within the home by a dietitian can increase energy, protein intake, and body weight. The goal of this study is to test a new model for continuity of nutrition care for malnutrition treatment across settings and determine if it improves food security and quality of life in patients 60 years and older. The study will specifically recruit sites and a sample that represents individuals who have malnutrition, have experienced or are at risk for food insecurity, and those from rural areas as well as Black, Latino, Indigenous and Native American populations with a goal sample size of 1,120 patients over the five-year duration. The objectives of this study are to: 1) test the feasibility of a patient identification, cross-referral, data reporting, and communication process from an acute care hospital to a community meal provision organization; 2) identify barriers to and facilitators for implementation as well as costs of the new model of continuity of nutrition care across settings; and 3) improve food security, determinants of malnutrition, and quality of life in persons older than 60 years of age discharged from the hospital with a diagnosis of malnutrition. Level 1 evidence will be generated from the study. The outcomes to be measured are program sustainability, percent change in referrals, food insecurity, malnutrition risk and diagnosis, and quality of life. The results of this study can provide a new model for nutrition care that may improve food security, quality of life, and health outcomes.

DETAILED DESCRIPTION:
We hypothesize that enhanced continuity of nutrition care between acute care hospital settings and community meal provision organizations providing Title III-C Special Need Plan services (C1 and C2) will be sustainable and improve outcomes for patients older than 60 years of age who are diagnosed with malnutrition. Specifically, the enhanced continuity of care will: a) increase referrals and communication between clinical and community nutrition care providers at each study site location; b) increase the percent of patients receiving nutrition care within the community setting; and c) improve food security, quality of life, and reduce determinants of malnutrition.

To test this hypothesis, we propose to conduct a study which will examine a new model of continuity of nutrition care for sustainability and impact. The model has been developed to facilitate cross-referrals and transmission of structured nutrition care documentation from an acute care setting to a meal provision organization and then for the meal provision organization to use the referral data to increase delivery of nutrition care (medical nutrition therapy- MNT) and meals (medically tailored meals - MTM). The primary subjects for this study are adults older than 60 years of age with malnutrition, with particular emphasis on recruiting sites who serve individuals who are Black, Latino, Indigenous and Native Americans and individuals living in rural areas of the country.

The components of the proposed new model of cross-referral, data transfer, and nutrition care across settings has the potential to be scalable throughout the US. However, barriers and facilitators to data transfer and MNT/MTM provision, cost of implementation, and potential impact on outcomes must be evaluated for the model to be replicable. The results of this study will generate new data on the model of care feasibility, rates of malnutrition within older adults at the study sites, impact of MNT with MTM provision on food security, determinants of malnutrition, and quality of life to inform future scalability of the model.

Goals and Objectives The goal of this new model is to improve food security and quality of life in patients 60 years and older from key vulnerable populations with greatest social and economic need by providing continuity of nutrition care for malnutrition treatment across settings. To test the feasibility of this new model, we will use a stepped wedge cluster-randomized trial design at eight sites throughout the US, specifically recruiting sites and individuals who are Black, Latino, Indigenous and Native American, and individuals living in rural areas of the country. The Academy of Nutrition and Dietetics (the Academy), as the research organization, and the Academy of Nutrition and Dietetics Foundation (Academy Foundation) will partner with collaborating organizations in both acute care hospitals and meal provision organizations (Title III-C1 and C2) within the community to test the newly developed model.

Objective 1) To test the feasibility of a patient identification, cross-referral, data reporting, and communication (including data transfer) process from an acute care hospital to a community meal provision organization.

Objective 1a) To identify barriers to and facilitators for implementation as well as the cost of the new model of continuity of nutrition care across settings.

Objective 2) To increase the rate of patients older than 60 years of age with malnutrition receiving care (MNT, MTM) in the community setting.

Objective 3) To improve food security, determinants of malnutrition, and quality of life in persons older than 60 years of age discharged from the hospital with a diagnosis of malnutrition.

There are two distinct portions of the study intervention: the clinical component, which includes patient identification, effective cross-referrals, and enhanced data reporting and transfer to the community partner, and the community component, including enhanced nutrition care and reporting including both MNT and MTM. The meals and nutrition care within the community can occur at home or within a congregate meal setting (Title III C1 and C2).

The study will compare the usual care process with no referral to the new model which includes a referral and nutrition care in the community using a stepped wedge cluster-randomized trial design.12 All participating sites will start in the control condition (usual process/care) and then be randomized to unidirectionally crossover to the intervention condition within four sequence blocks on a staggered schedule (see work plan year 2 for detailed table). Patients diagnosed with malnutrition in the hospital setting will be cross-sectionally identified and enrolled within each study period. All enrolled patients, regardless of whether they are in the control or receive the intervention will have outcome measures collected 3 months post-discharge (+/- two weeks). All sites will begin in the control period and then two sites at a time will implement the intervention in a staggered approach. Thus, in period 1 all are following usual care, then in period 2, two sites will implement the new model, in period 3, two additional sites will implement it, and this will continue until all sites have implemented the new model (intervention) at the end of period 5. Each period will last 7 months for a total study duration of 35 months. Patient recruitment will occur within all 5 periods for a total of 1120 patients and at a rate of approximately six to seven patients per month per site. This approach ensures all sites test the intervention and evaluate sustainability and impact of the new model.

Clinical setting: Standards for usual care within the hospital includes screening for malnutrition risk by nursing or other non-RDN staff, 14 within 24 hours of admission. A positive screening elicits a consultation with an RDN who conducts a comprehensive assessment to determine whether a nutrition problem, such as malnutrition, exists. The RDN will then provide nutrition care to patients for the duration of their hospital stay. The nutrition care is documented in the hospital's electronic health record (EHR) and includes anthropometric and laboratory data in addition to the nutrition problem and care plan.For the new model of care, the data collection tool (ANDHII) will be modified to use the HL7® FHIR standard to import (pull) data from acute care hospital EHRs. The data will then be available via ANDHII for the community RDN to use.

Community setting: Within our new model of continuity of nutrition care, an RDN within the meal provision organization (Title III-C1 and 2) will log into ANDHII and accept the referral and subsequent data sent by the clinical RDN. The community RDN will review the data and the discharge nutrition care plan before visiting with the patient within their home or at the congregate meal center. At the initial community visit (home visit or congregate meal site), the community RDN will reassess the person for malnutrition and adjust the nutrition care plan as needed for the home/community environment and the patient's social, functional, and economic circumstances. The aim within the community setting will be for the community RDN to have three subsequent visits, approximately a month apart, for three months post-discharge from the hospital. A dedicated Research RDN at each site will conduct the malnutrition, food security, and QOL tools at baseline and again at the end of month three post-discharge for all the enrolled patients, regardless of whether they are in the control or intervention period.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking,
* Screened as at risk for malnutrition (Malnutrition Screening Tool),
* Meet the definition for food insecure per the Food Security Risk tool,
* Referred to an RDN,
* Diagnosed with malnutrition using AAIM,
* Plan for discharge to home, and
* Eligible to receive Title III-C1 or Title III-C2 nutrition services.

Exclusion Criteria:

* Patients are receiving hospice care or care for end stage cancer,
* Unable to consume meals (e.g., using enteral or parenteral to meet nutrition needs), Do not live within the meal provision organizations catchment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale (CASP-19) | 3 months
  This tool has been validated in older populations and examined in populations with lower socioeconomic status and in different racial and ethnic populations. It will be conducted to evaluate the change in quality of life over time as a result of the intervention.

SECONDARY OUTCOMES:
Program Sustainability Assessment Tool | Facility level outcome, thus outcome will be done at study completion for the site years 2 through 4
  The Program Sustainability Assessment Tool (PSAT) is based on a sustainability framework with eight domains (environmental support, financial stability, communications, strategic planning, partnerships, program adaptation, program evaluation, organizational capacity). Each of these domains provides insight into the program's sustainability and opportunities for enhancement. The assessment tool has 40 questions within the eight domains and will be completed by the research RDN. It takes approximately 10-15 mins to complete and thus has minimal staff burden.
RDN Survey on Barriers and Facilitators to Implementation | Facility level outcome, thus outcome will be done at study completion for the site years 2 through 4
  A survey which has been developed and used within Academy research projects, will be modified to assess this new model.
Change in percent of patients receiving nutrition care and meals | 3 months
  Pre and post numbers of patients who have malnutrition and are referred from the acute care setting to the community setting receiving care by an RDN and meals from meal provision title III-C1 and C2 funded organizations will be captured and calculated for a percent change from the control period to post implementation of the new model
Food Security Risk | 3 months post discharge from the hospital
  The food security risk assessment tool is valid has 6 questions and will be used to determine security risk.
Malnutrition risk | baseline in hospital and at 3 months post discharge from the hospital
  The malnutrition screening tool is a valid tool for determining risk of malnutrition in adults.
Malnutrition Diagnosis (AAIM tool) | 3 months post discharge from the hospital
  Validated diagnostic tool for moderate and severe malnutrition in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Alison L Steiber, Principal Investigator — Academy of Nutrition and Dietetics

IPD SHARING:
Plan to Share IPD: No